CLINICAL TRIAL: NCT00195026
Title: Infrared Imaging (Breast Scan IR) for Early Breast Cancer Detection
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Dr. Rache Simmons, Weill Cornell Medical College
Other Study IDs: 0309006370
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Last update posted 2008-03-18 (Estimated); Status verified 2008-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Device: Infrared Breast Scan — Patients already scheduled for breast biopsies will receive an additional infrared scan

SUMMARY:
This protocol will evaluate a new non-invasive infrared imaging system as an adjunctive tool for breast cancer detection that has been approved by the FDA. The technology and device have been developed by Infrared Sciences Corp. and has undergone more than 3 years of testing prior. The subject device's utility will be investigated with regard to its sensitivity toward breast cancer, however it records temperature data and other physiological parameters of the breast, and compares them to a database of patients with known breast health.

DETAILED DESCRIPTION:
The research study will evaluate the sensitivity and specificity of a new non-invasive digital infrared imaging system as an adjunctive test for breast cancer detection (as approved by the FDA under 21 CFR 884.2980). The technology and device (BreastScan IRÔ) have been developed by Infrared Sciences Corp. and has undergone more than 3 years of preliminary testing. The device's utility will be investigated with regard to its sensitivity in detecting breast cancer, and its ability to identify the size of the breast cancer. Additionally, the negative predictive value of the device will be investigated. This device does not diagnose breast cancer, however it records temperature data and other physiological parameters of the breast, and compares them to a database of patients with known breast health.

The examination process is simple and non-invasive. The patient sits disrobed from the waist up, appropriately positioned in the ergonomic chair with her arms supported at eye level. Temperature controlled air flow is then directed at the breasts for a 4-minute interval while the infrared camera records skin surface cool down at 250 frames per minute. The stored images are fed into proprietary computer software designed to extract specific thermal parameters, including various temperature differences and thermal symmetry measurements. Additionally, the software will focus on areas of the breasts, when compared to its immediate surroundings, that behave abnormally. The program produces a color coded post-processed image of the breasts showing one or more these identified sites, as well as the result of all measured parameters. The combination of these parameters are evaluated for risk in a weighted "evaluation" algorithm, as determined by the information in the database. The results of the digital infrared scan will be correlated with the results of the subsequent breast biopsy.

Selected patients will be required to sign an informed consent form. These patients will have been recommended to have a biopsy, based either on mammography or ultrasound. The patients overall breast density will be noted. Each patient will be "imaged" with the BreastScan IR system, and the raw data stored. The computer will analyze the raw data, and will produce a report showing the results of the test. This report will be stored for use once the results of the patient's biopsy is known.

For each patient, the report will provide an evaluation of "risk" as well as other data that will help localize any suspicious sites. Comparison will be made with actual radiology and pathology results.

If a patient is determined by biopsy to have any form or breast cancer, or atypical hyperplasia, the investigator will examine the BreastScan IR report, and verify that this patient was evaluated as "Risk" (one or more positive risk signs). If sufficient information is provided in the pathology or radiology report to determine the site(s) in the breast, the investigator will again verify that the BreastScan IR report correctly localizes the breast and quadrant of the known cancer. The incidence of incorrect evaluations will be recorded for determination of the system's sensitivity to breast cancer.

If a patient is determined by biopsy to have any non-malignant condition, such as a cyst or fibroadenoma, the investigator will determine if the BreastScan IR report evaluated the patient as "Normal" (zero positive signs) or as "Risk".

Methodology:

Two hundred (200) female patients will be selected from a normal screening process. Those patients that have a finding that is suspicious for cancer (BIRADS 3) or highly suspicious for cancer (BIRADS 4,5), and/or that have been scheduled for a biopsy, will be included in this study. The patients will be asked to sign an informed consent form.

Data:

The data collected in this trial will be blinded to the patient as well as the radiologist. The data for an individual patient will be stored locally, within the BreastScan IR system, and will not be available to anyone except authorized research investigators. The data will be stored for future use and analysis. Since this data must be compared to an actual radiology/pathology report, the data cannot be anonymous, but will be confidential.

Patient Risk:

The test is completely non-invasive, and presents no risk whatsoever to the patient. The infrared camera records infrared energy emitted from the patient's body. Cool air is not excessively cold, and does not present any discomfort to most patients.

Benefits:

The main objective of the test is to develop a tool that will help diagnose breast cancer by providing accurate adjunctive information to the patient's doctor. Preliminary studies indicate that this test is 99% sensitive to breast cancer. A patient with a "normal" (negative) result will have a very small chance that an occult cancer is still harbored in the breast. Conversely, a patient that has an abnormal test will require further work-up.

We hope to benefit two groups of women that now account for largest proportion of "missed" cancers. Namely, those women with dense breast tissue, and those women under 40 who are at the pre-mammography age, and who generally have dense breast tissue. A non-invasive test that can help with improved screening, is urgently needed to improve the detection statistics in these groups, and hopefully lead to early intervention of those patients at high risk.

ELIGIBILITY:
Inclusion Criteria:

* Mammographic Breast Abnormality requiring a follow up biopsy
* Sonographic Breast Abnormality requiring a follow up biopsy
* Clinical Breast Abnormality requiring a follow up biopsy

Exclusion Criteria:

* Active Breast Inflammation
* Previous history of breast augmentation
* Bra size greater than DD

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients already recommended for breast biopsy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2005-03

CONTACTS AND LOCATIONS:
Overall Officials: Michael Osborne, MD, Principal Investigator — NY Presbyterian Hospital Weill Cornell Breast Center
Locations (1):
- Weill Cornell Breast Center, New York, New York, United States